CLINICAL TRIAL: NCT01596829
Title: Effect of Probiotic Formula on Reducing the Risk for Antibiotic-associated Diarrhoea
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low incidence
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AAD-EU2012; 2012-001542-18 (EudraCT Number)
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2014-12

CONDITIONS: Antibiotic-associated Diarrhoea
Keywords: antibiotic; probiotic; antibiotic-associated diarrhoea; faecal microbiota
MeSH Terms: interventions — Probiotics; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic consumption during and after course of antibiotic
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo consumed during and after course of antibiotic
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic formula, 10 billion CFU in total once a day for up to 3 weeks
  Other Names: Howaru Restore
  Arms: Probiotic
Dietary Supplement: Placebo — A capsule with microcrystalline cellulose matching the appearance and taste of the active comparator
  Other Names: Microcrystalline cellulose as placebo
  Arms: Placebo

SUMMARY:
Antibiotic treatment disturbs the balance of the intestinal microbiota and predisposes to antibiotic associated diarrhea. Previous studies have shown that the risk of developing diarrhea during a course of antibiotics may be reduced by simultaneous consumption of probiotics. The aim of the present study is to assess the effect of a probiotic formula containing four strains on reducing the risk of antibiotic associated diarrhea.

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of a probiotic formula on reducing the risk of antibiotic-associated diarrhea (AAD). The study will be conducted as a two-arm, parallel groups, placebo-controlled, double-blind, randomized clinical trial, stratified by age, gender and number of days on antibiotics. The duration of patient participation in the study will be up to 7 weeks (up to 3 weeks supplementation, 4 weeks follow-up). The overall duration of the study is expected to be approximately 8 months. Adult males and females that are prescribed antibiotic therapy for minimum of 3 and a maximum of 14 days will be included in the study. The incidence of AAD will be evaluated as the primary end-point. The stool from patients presenting diarrhea will be tested for the presence of Clostridium difficile and if negative for C. difficile, also for the presence of other common pathogens causing diarrhea. The overall microbiota will be analyzed from fecal samples taken regularly during each phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-65 years.
2. Patients will be initiating antibiotic therapy.
3. The antibiotic therapy consists of one of the following: broad spectrum penicillins, cephalosporins, doxycycline, clarithromycin, ciprofloxacin or isoxazolyl penicillin.
4. The antibiotic therapy is expected to be 3 to 14 days in duration.
5. Obtained his/her informed consent after verbal and written information.
6. Have a high probability for compliance with and completion of the study.
7. Patients having a telephone available.
8. Body Mass Index between 19 and 30.

Exclusion Criteria:

1. Participation in a clinical trial with an investigational product or drug within the 60 days prior to screening.
2. Likeliness to be noncompliant with the protocol, or to be unsuitable to the study by the investigator for any reason.
3. Pregnant or breastfeeding women; women planning to become pregnant during the study months.
4. Presence of active diarrhea (3 or more loose or watery stools per 24 hour period).
5. Daily consumption of probiotics, fermented milk and/or yogurt with probiotics.
6. Known to have a previous reaction, including anaphylaxis, to any substance in composition of the study product (i.e. on-medicinal ingredients: Cellulose, hypromellose, magnesium stearate (vegetable source), ascorbic acid, Colloidal silicon dioxide).
7. Presence of an active, non-controlled intestinal disease such as Crohn's Disease or ulcerative colitis.
8. Regular use of proton pump inhibitors.
9. Bowel surgery, artificial heart valve, history of rheumatic heart disease or infective endocarditis.
10. A previous documented C. difficile infection < 3 months prior to study initiation.
11. Immunosuppressive therapy or any health condition causing immunosuppression (including haematological malignancies, AIDS).
12. Ongoing or recent use of antibiotic therapy in the 3 months prior to the study product first administration.
13. Planned administration of antibiotics other than broad spectrum penicillins, cephalosporins, doxycycline, ciprofloxacin or isoxazolyl penicillin for the treatment of an infection.
14. History of drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AAD | Up to 21 days
  Incidence of diarrhoea defined as three or more loose or watery stools per a 24 h period.

SECONDARY OUTCOMES:
Duration of diarrhoea | Up to 21 days
  Number of continuous days of diarrhoea
Fecal microbiota | Up to 21 days
  Analysis of overall microbiota from all samples and of causative diarrhoeal agent from samples taken during diarrhoeal episode
Safety profile | Up to 21 days
  Evaluation of serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Toivo Piippo, MD, Principal Investigator — Koskiklinikka Tampereen Lääkärikeskus Oy; Anneli Tarpila, PhD, Study Chair — Danisco
Locations (1):
- Koskiklinikka, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No
Terminated prematurely.

REFERENCES:
- [Derived] Forssten SD, Yeung N, Ouwehand AC. Fecal Recovery of Probiotics Administered as a Multi-Strain Formulation during Antibiotic Treatment. Biomedicines. 2020 Apr 9;8(4):83. doi: 10.3390/biomedicines8040083. PMID 32283645